CLINICAL TRIAL: NCT02988258
Title: CMV TCR Gene Therapy: A Phase I Safety, Toxicity and Feasibility Study of Adoptive Immunotherapy With CMV TCR-transduced Donor-derived T Cells for Recipients of Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Study of Adoptive Immunotherapy With Donor-derived CMV-specific T Cells for Recipients of Allo-HSCT
Acronym: CMV_TCR-001
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol being re-written to allow inclusion of more patients
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL 08/0214; 2008-006649-18 (EudraCT Number); G0701703 (Other Grant/Funding Number: Medical Research Council (MRC)); 08/0214 (Other: Sponsor Number)
Record Dates: First submitted 2012-07-12; First posted 2016-12-09 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Haematological Malignancies; CMV Infection
Keywords: Ex vivo gene therapy; T cell receptor transduction; Immunotherapy; Allogeneic Haematopoietic Stem Cell Transplantation; CMV
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 - 10^4 transduced cells/kg (Experimental): The first 3 patients will receive a single infusion of bulk CMV-TCR transduced donor-derived T cells on first CMV reactivation post allogeneic HSCT, at a dose of 10^4 T cells/kg recipient weight
  Interventions: Genetic: CMV-TCR transduced donor-derived T cells
- Cohort 2 - 10^5 transduced cells/kg (Experimental): If no cases grade III-IV GVHD in Cohort 1 the remaining patients (N=7) each receive a single infusion of bulk CMV-TCR transduced donor-derived T cells on first CMV reactivation post allogeneic HSCT, at a dose of 10^5 T cells/kg recipient weight
  Interventions: Genetic: CMV-TCR transduced donor-derived T cells
- Cohort 1a - 10^3 transduced cells/kg (Experimental): If 1 case grade III-IV GVHD in Cohort 1, next three patients to be treated with a single infusion of bulk CMV-TCR transduced donor-derived T cells of 1 x 10^3 T cells/kg recipient weight
  Interventions: Genetic: CMV-TCR transduced donor-derived T cells

INTERVENTIONS:
Genetic: CMV-TCR transduced donor-derived T cells — Dose escalation

SUMMARY:
The study will test the hypothesis that CMV TCR-transduced T cells, at a specific T-cell dose/kg, can generate a functional CMV immune response post-transplant, where CMV-specific donor T cells cannot be isolated by conventional means. This will be tested in the context of adult HLA-matched sibling allogeneic HSCT.

In the proposed trial, an HLA-A*0201-restricted CMV pp65-specific T cell receptor (TCR) will be introduced into donor T cells via ex vivo GMP retroviral transduction. Donor T cells will be isolated from peripheral blood following a simple venesection procedure. The CMV TCR-transduced T cells will be tested for TCR expression, CMV-specific cytokine secretion and microbiological contamination before being frozen and stored at -80C. CMV seropositive transplant recipients will be tested weekly for CMV reactivation by quantitative PCR on peripheral blood. On first detection of CMV DNA > 200 copies/ml, 104 (cohort 1) or 105 (cohort 2) bulk CMV TCR-transduced T cells/kg recipient weight will be infused into the patient.

Blood will be taken regularly to determine persistence and expansion of the CMV TCR-transduced T cells. Weekly CMV PCR will be continued. Patients will be examined at appropriate intervals (daily if inpatients, twice weekly in BMT clinic if outpatients) for the development of graft versus host disease (GVHD) or other potential side effects.

DETAILED DESCRIPTION:
Reactivation of the latent human herpes virus, Cytomegalovirus (CMV), post allogeneic haematopoietic stem cell transplantation (Allo-HSCT) can result in significant morbidity and mortality unless treated promptly. Anti-viral therapy is usually effective, but has serious side effects typically requiring prolonged inpatient admission, such as myelosuppression (Ganciclovir) or nephrotoxicity (Foscarnet). Cellular immunotherapy for CMV has been tested in Phase I/II trials in the UK and Europe. In these trials CMV-specific T cells were isolated from the peripheral blood of CMV seropositive donors and re-infused into recipients following CMV reactivation resulting in sustained anti-viral responses. It is clear that post-transplant recovery of CD8+ CMV-specific cytotoxic T-cells (CTL) abrogates the development of CMV-related disease. An advantage of cellular therapy for CMV reactivation is the transfer of immunological memory, which can reduce the number of subsequent reactivations. This is important, as rapidly increasing numbers of highly immunosuppressive (or T cell depleted) reduced intensity conditioning Allo-HSCTs are being performed in the UK. These approaches reduce the toxicity of transplantation in older patients with more co-morbidities. Reduced intensity allogeneic transplants are currently part of the UK MRC AML15 trial and are to be recommended in the proposed MRC/ECOG UKALL14 study and again in UK MRC AML17. In addition, a number of NCRN approved UK multicentre extended Phase II studies have recently started using reduced intensity Allo-HSCT in various lymphoma subtypes.

Transplant recipients with CMV seronegative donors cannot benefit from currently available cellular immunotherapy approaches due to the lack of CMV-specific memory T cells in these donors. At present, there is no reliable strategy to isolate virus specific T cells from uninfected naïve individuals, as the precursor frequency is low or absent and the in vitro priming of T-cell responses is inefficient. T-cell receptor (TCR) gene transfer offers a strategy to produce antigen-specific T cells independent of precursor frequency and without the need for T-cell priming. As approximately 50% of adult individuals have been previously infected with CMV, there are significant numbers of CMV 'mismatched' Allo-HSCT performed, where the donor is CMV seronegative and the recipient CMV seropositive. The proposed study will test the feasibility of generating donor-derived CMV-specific T cells via the ex vivo introduction of a CMV-specific T cell receptor using a GMP grade retroviral vector.

ELIGIBILITY:
Patient Inclusion Criteria:

* Undergoing matched sibling allogeneic HSCT for an underlying haematological malignancy with a CMV seronegative donor
* Age ≥ 18 years and ≤ 65 years
* HLA-A*0201 positive
* CMV seropositive (CMV IgG detected) pre-transplant
* Informed consent in writing and ability to co-operate with treatment and follow up.

  * Prepared to undergo additional study procedures as per study schedule
  * Patient has undergone counselling about risk
* Serologically negative for HIV 1&2, Hep B, Hep C and syphilis
* Female patients of child-bearing age must have a negative pregnancy test and agree to use reliable contraceptive methods for the duration of the therapy and for 6 months afterwards
* Male patients must agree to use appropriate medically approved contraception during the trial and for six months afterwards

And to be assessed prior to CMV-specific T cell infusion (for confirmation prior to product release):

* Donor engraftment (neutrophils > 0.5x109/l).
* Single positive CMV PCR result (> 200 copies/ml)

Patient Exclusion Criteria:

* Pregnant or lactating women
* Co-existing medical problems that would place the patient at significant risk of death due to GVHD or its sequelae
* HIV infection

And to be assessed prior to CMV-specific T cell infusion (for confirmation prior to product release):

* Active acute GVHD > Grade I
* Concurrent use of systemic corticosteroids
* Organ dysfunction as measured by

  * creatinine > 200 uM/l
  * bilirubin > 50 uM/l
  * ALT > 3x upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-07; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Determination of the frequency of transduced donor-derived cells expressing the CMV-specific TCR by flow cytometry. | 5 years
  CMV-TCR transduced cells express vbeta13 and murine constant beta chain (mCb), both of which can be easily detected by flow cytometry. The frequency of vbeta13+/mCb+ is used to calculate the efficiency of transduction of donor-derived cells.
Evaluation of treatment toxicity according to the NCI Common Toxicity Criteria Scale (v4.03). | 5 years

SECONDARY OUTCOMES:
Documentation of anti-CMV responses post CMV-TCR transduced cell infusion using quantitative PCR to determine viral copy numbers in peripheral blood. | 5 years
Evaluation of GvHD post CMV-TCR transduced cell infusion following allo-HSCT using standardised international criteria. | 5 years
Evaluation of immune reconstitution post CMV-TCR transduced cell infusion following allo-HSCT. | 5 years
  Flow cytometry and TCR repertoire analysis can be used to evaluate overall T-cell subset reconstitution.
Assessment of the number of CMV-TCR transduced cells that are able to persist post-infusion using quantitative real-time PCR. | 5 years
  Quantitative real-time PCR using primers specifically targeting nucleotide sequences that are only present in the introduced CMV-TCR can be used to determine the number of circulating CMV-TCR transduced cells post infusion.
Phenotypic characterisation of CMV-TCR transduced cells by flow cytometry in terms of relative expression of markers associated with cell differentiation, proliferation and intracellular cytokine production. | 5 years
  Flow cytometry can be used to further characterise CMV-TCR transduced cells in terms of naive/memory subsets (based on the expression of CD45RO and CD62L differentiation markers), proliferation status (assessed by Ki-67) and ability to produce cytokines (such as IFN-gamma and TNF-alpha).

CONTACTS AND LOCATIONS:
Overall Officials: Emma Morris, Prof, Principal Investigator — University College, London; Hans Stauss, Prof, Study Chair — University College, London
Locations (4):
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University College London Hospital, London
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tendeiro Rego R, Morris EC, Lowdell MW. T-cell receptor gene-modified cells: past promises, present methodologies and future challenges. Cytotherapy. 2019 Mar;21(3):341-357. doi: 10.1016/j.jcyt.2018.12.002. Epub 2019 Jan 14. PMID 30655164